CLINICAL TRIAL: NCT00907140
Title: Assessment of Changes in Pattern and Magnitude of Tumor FDG Uptake During Chemoradiation as a Predictor of Response to Concurrent Radiation Therapy and Chemotherapy in Patients With Cervical Cancer
Brief Title: Fludeoxyglucose (FDG) Positron Emission Tomography/Computed Tomography (PET/CT) Cervical Heterogenity Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Farrokh Dehdashti, Co-Principal Investigator, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-0804
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Positron Emission Tomography; Fluorodeoxyglucose
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiation therapy (Other)
  Interventions: Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Positron Emission Tomography — FDG PET/CT imaging is performed at baseline, after 2 and 4 weeks of radiation therapy and approximately 3 months after chemoradiation is completed

SUMMARY:
Rationale: Diagnostic procedures, such as positron emission tomography (PET) using fluorodeoxyglucose (FDG), may help determine response to standard cancer therapy in patients with cervical cancer

The purpose of this study is to evaluate the change in cervical tumor heterogenity as measured by FDG-PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven cervical cancer. (FIGO stage-Ib2-IVa)
2. Age ≥ 18
3. Able to receive chemoradiation therapy with Cisplatin.
4. Non-pregnant status in women of childbearing potential.
5. No other active cancer at the time of diagnosis of cervical cancer Patients cannot have received treatment for any malignancy, with the exception of non-melanoma skin cancer, in the past 5 years.
6. Patients with distant metastatic disease are eligible provided the estimated survival of the patient is at least 1 year.
7. Scheduled to undergo or have already undergone FDG-PET/CT imaging for clinical staging of cervical cancer at Barnes-Jewish Hospital Clinical PET Facility on a Biograph 40 PET/CT scanner
8. Able to give informed consent

Exclusion Criteria:

1. Age < 18
2. Patients with a known active malignancy other than cervical carcinoma.
3. Pregnant and breastfeeding patients.
4. Subjects whose tumors are not FDG avid on baseline standard of care FDG-PET/CT imaging

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The overall goal of this pilot study is to evaluate the change in cervical tumor FDG heterogeneity and SUVmax during chemoradiation. | FDG PET/CT imaging is performed at: Baseline, 2 & 4 weeks of therapy, and 3 months after completing therapy

SECONDARY OUTCOMES:
To correlate changed in FDG heterogeneity and SUVmax with response to therapy. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Perry W Grigsby, M.D., Principal Investigator — Washington University at St. Louis
Locations (1):
- Washington University at St. Louis, St Louis, Missouri, United States